CLINICAL TRIAL: NCT00571740
Title: Randomized Phase II Trial of Cetuximab/Bevacizumab (CB) as Palliative First-Line Therapy in Patients With Advanced Colorectal Cancer Followed by FOLFOX+CB vs. FOLFOX+B
Brief Title: Cetuximab and Bevacizumab as First-Line Therapy Followed By Combination Chemotherapy and Bevacizumab With or Without Cetuximab as Second-Line Therapy in Treating Patients With Stage IV Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not activated
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0548; CDR0000578111 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00651 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Leucovorin; Oxaliplatin

ARMS (2):
- Arm I (second-line therapy) (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- Arm II (second-line therapy) (Experimental): Patients receive bevacizumab and modified FOLFOX7 as in arm I. Patients also receive cetuximab IV over 2 hours on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Biological: cetuximab; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
Biological: cetuximab — Given IV
  Arms: Arm II (second-line therapy)
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving monoclonal antibodies together with combination chemotherapy may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving cetuximab together bevacizumab works as first-line therapy, followed by combination chemotherapy and bevacizumab with or without cetuximab as second-line therapy in treating patients with stage IV colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy of bevacizumab and cetuximab as first-line treatment for metastatic colorectal cancer, as measured by percentage of patients who remain progression-free at 6 months.

Secondary

* To evaluate adverse events, confirmed response, duration of response, time to disease progression, time to treatment failure, and survival of patients treated with bevacizumab and cetuximab.
* To evaluate adverse events, confirmed response, duration of response, time to disease progression, time to treatment failure, and survival of patients who are refractory to dual-agent bevacizumab and cetuximab and are subsequently treated with modified FOLFOX7 chemotherapy and bevacizumab with or without cetuximab.
* To evaluate quality of life parameters in patients treated with these regimens.
* To estimate the direct medical resource utilization and costs.
* To assess the reliability of FDG-PET as a measurement of early treatment response, as measured by percentage of patients who are progression-free at 6 months.
* To identify circulating angiogenesis biomarkers.
* To assay the activity of pro-angiogenic factors in plasma angiogenic assays.

OUTLINE: This is a multicenter study*. Patients are stratified according to ECOG performance status (0-1 vs 2) and number of metastatic sites (1 vs > 1).

NOTE: *Participating site must be PET-qualified.

* First-line therapy: Patients receive bevacizumab IV over 30-90 minutes and cetuximab IV over 2 hours on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients with progressive disease proceed to second-line therapy.
* Second-line therapy: Patients are randomized* to 1 of 2 treatment arms.

  * Arm I (modified FOLFOX7 with bevacizumab only): Patients receive bevacizumab IV over 30-90 minutes, oxaliplatin IV over 2 hours, and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV over 46 hours beginning on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.
  * Arm II (modified FOLFOX7 with bevacizumab and cetuximab): Patients receive bevacizumab and modified FOLFOX7 as in arm I. Patients also receive cetuximab IV over 2 hours on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *Randomization occurs prior to receiving first-line therapy.

Patients undergo blood sample collection periodically for translational studies. Samples are analyzed for circulating endothelial cells and endothelial progenitor cells via flow cytometry; angiogenic activity of serum/plasma in angiogenesis-dependent diseases via endothelial proliferation assay and matrigel tube formation assay; and circulating angiogenesis biomarkers (i.e., free VEGF, soluble FLT-1, and KDR) via ELISA.

Quality of life is assessed periodically using the UNISCALE, Skindex-16, and Skin Assessment Questionnaires.

After completion of study treatment, patients are followed every 6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV colorectal cancer
* Measurable disease, defined as at least one lesion whose longest diameter can be accurately measured as ≥ 2.0 cm by conventional techniques OR ≥ 1.0 cm by spiral CT scan
* Must not be a candidate for neoadjuvant therapy
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN
* AST ≤ 3 times ULN
* Creatinine ≤ 1.5 x times ULN
* Proteinuria < 1+ by urinalysis OR proteinuria < 1 g by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* English-speaking patients must have the ability to complete questionnaires by themselves or with assistance
* Must be willing to provide blood and tissue samples for research purposes
* No history of hypertensive crisis or hypertensive encephalopathy
* No blood pressure > 150/100 mm Hg
* No New York Heart Association (NYHA) class II-IV congestive heart failure
* No myocardial infarction or unstable angina within the past 6 months
* No stroke or transient ischemic attack within the past 6 months
* No clinically significant vascular disease (e.g., aortic aneurysm or aortic dissection)
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 28 days
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious nonhealing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

* No prior nonsurgical treatment for stage IV disease

  * Adjuvant therapy allowed if completed > 6 months prior to study registration
* More than 4 weeks since prior and no concurrent or planned participation in another experimental drug study
* No prior therapy that specifically and directly targets the EGFR pathway
* No prior monoclonal antibody therapy
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior minor surgery, such as fine-needle aspirations or core biopsies

  * Placement of a vascular access device does not have to meet this criterion
* No concurrent major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 6 months | at 6 months

SECONDARY OUTCOMES:
Tumor response rate associated with second-line therapy | up to 3 years
Time to progression during second-line therapy | up to 3 years
Duration of response | up to 3 years
Quality of life | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Axel Grothey, MD, Study Chair — Mayo Clinic